CLINICAL TRIAL: NCT00797628
Title: QUIT-PRIMO: Web-Delivered Clinical Microsystem Intervention for Tobacco Control
Brief Title: Web-delivered Provider Intervention for Tobacco Control
Acronym: QUIT-PRIMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Johns Hopkins University (Other); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Thomas Houston, Principal Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: X071211009; NIH R01CA129091
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Information Prescription (Experimental): Providers will give usual care to patients who smoke and a paper prescription with the name and url of the "Smoking Coach" website. The smoking coach website is a tailored, public health intervention for smoking cessation.
  Interventions: Behavioral: Smoking Coach
- QUIT-PRIMO (Experimental): Providers will give usual care to patients who smoke and then refer patients to the online smoking cessation system electronically.
  Interventions: Behavioral: Decide2Quit

INTERVENTIONS:
Behavioral: Decide2Quit — Patient intervention website that includes 1) interactive calculators to assess readiness to quit, symptoms and quit plan, 2) motivational content, and 3) links to other high quality information.
  Arms: QUIT-PRIMO
Behavioral: Smoking Coach — Control Patients will be referred by paper prescription to the control- "Smoking Coach" website.
  Arms: Information Prescription

SUMMARY:
This is a randomized control trial to determine the efficacy of a multi-modal intervention in improving smoking cessation processes of care and patient outcomes in community-based primary care practices. Our Overall Goal is to advance science related to the use and impact of the Internet in health services delivery, specifically smoking cessation, by targeting primary care clinical microsystems. A clinical microsystem is defined as the smallest functional healthcare unit. A clinical microsystem is not simply equivalent to a clinical team of doctors and nurses, but also the panel of patients cared for by the providers and the processes of care that are used.

ELIGIBILITY:
Inclusion Criteria:

* Community based primary care practices who have:

  * Internet access in office
  * Sees 4 - 5 smokers per week

Exclusion Criteria:

* Practices with more than five providers

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2010-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Physician performance on refering patients that smoke cigarettes to the web intervention | pre-intervention, 6 months, 12 months and 24 months
Of the smokers who are referred to the web intervention, the number who go to the site | preintervention, 6 months, 12 months, 24 months
Point prevalence smoking cessation | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas K Houston, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

REFERENCES:
- [Derived] DeLaughter KL, Sadasivam RS, Kamberi A, English TM, Seward GL, Chan SW, Volkman JE, Amante DJ, Houston TK. Crave-Out: A Distraction/Motivation Mobile Game to Assist in Smoking Cessation. JMIR Serious Games. 2016 May 26;4(1):e3. doi: 10.2196/games.4566. PMID 27229772
- [Derived] Houston TK, Sadasivam RS, Allison JJ, Ash AS, Ray MN, English TM, Hogan TP, Ford DE. Evaluating the QUIT-PRIMO clinical practice ePortal to increase smoker engagement with online cessation interventions: a national hybrid type 2 implementation study. Implement Sci. 2015 Nov 2;10:154. doi: 10.1186/s13012-015-0336-8. PMID 26525410
- [Derived] Coley HL, Sadasivam RS, Williams JH, Volkman JE, Schoenberger YM, Kohler CL, Sobko H, Ray MN, Allison JJ, Ford DE, Gilbert GH, Houston TK; National Dental PBRN and QUITPRIMO Collaborative Group. Crowdsourced peer- versus expert-written smoking-cessation messages. Am J Prev Med. 2013 Nov;45(5):543-50. doi: 10.1016/j.amepre.2013.07.004. PMID 24139766
- [Derived] Sadasivam RS, Kinney RL, Delaughter K, Rao SR, Williams JH, Coley HL, Ray MN, Gilbert GH, Allison JJ, Ford DE, Houston TK; National Dental PBRN Group; QUIT-PRIMO Collaborative Group. Who participates in Web-assisted tobacco interventions? The QUIT-PRIMO and National Dental Practice-Based Research Network Hi-Quit studies. J Med Internet Res. 2013 May 1;15(5):e77. doi: 10.2196/jmir.2385. PMID 23635417
- [Derived] Sadasivam RS, Delaughter K, Crenshaw K, Sobko HJ, Williams JH, Coley HL, Ray MN, Ford DE, Allison JJ, Houston TK. Development of an interactive, Web-delivered system to increase provider-patient engagement in smoking cessation. J Med Internet Res. 2011 Oct 18;13(4):e87. doi: 10.2196/jmir.1721. PMID 22011394
- [Derived] Houston TK, Sadasivam RS, Ford DE, Richman J, Ray MN, Allison JJ. The QUIT-PRIMO provider-patient Internet-delivered smoking cessation referral intervention: a cluster-randomized comparative effectiveness trial: study protocol. Implement Sci. 2010 Nov 17;5:87. doi: 10.1186/1748-5908-5-87. PMID 21080972